CLINICAL TRIAL: NCT04044820
Title: Discharge Opioid Prescription for Ambulatory Hand and Forearm Surgery: A Randomized Controlled Trial
Brief Title: Opioid Use Post-Discharge After Ambulatory Distal Arm Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-5539
Record Dates: First submitted 2019-05-23; First posted 2019-08-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Discharge Prescription (Active Comparator): Based on a previous study examining mean number of opioid pills used by patients undergoing elective, unilateral hand and forearm surgery
  Interventions: Drug: Standardized Prescription
- Usual Discharge Prescription (No Intervention): Routine standard of care involves prescription for opioids at the discretion of the surgical team

INTERVENTIONS:
Drug: Standardized Prescription — Oxycodone 5mg PO q4-6h PRN
  If patient has allergy or other contraindications
  Hydromorphone 1mg PO q4-6h PRN/ Tylenol #3 1-2 tablets PO q4h PRN
  The number of tablets prescribed will depend on the extent of surgical trauma
  * 0-5 pills for simple surgeries such as a trigger finger release
  * 10 pills for carpal tunnel or Dupuytren's contracture releases
  * 15 pills for a ganglion cyst excision or simple tendon transfer
  * 20 pills for more complex procedures such as distal forearm ORIF or a wrist fusion.
  Arms: Standardized Discharge Prescription

SUMMARY:
The aim of this study is to determine if a standardized evidence-based opioid prescription following elective hand and forearm surgery at Toronto Western Hospital (TWH) will decrease the number of unused opioid pills consumed by patients while still maintaining adequate pain control as compared to usual treatment. Currently, no standardized prescription exists at our institution.

DETAILED DESCRIPTION:
This study is a Prospective Randomized Controlled Trial with an aim to determine if a standardized discharge prescription provides effective analgesia while reducing the number of unused opioid pills in the community.

All patients presenting to TWH during the recruitment phase for elective ambulatory hand and arm surgery will be asked to participate in the study. Patients will be given information about the study in the pre-operative surgical clinic by the surgeon assessing them. If agreeable, patients will then be approached for recruitment by a research assistant.

Patients would be randomized to either standardized prescription arm versus control arm (usual prescriptions administered by physician).

The standardized prescription will consist of an opioid prescription for Oxycodone 5mg PO q4-6h PRN. Alternatively, if the patient has an allergy or other contraindication to Oxycodone, Hydromorphone 1mg PO q4-6h PRN or Tylenol #3 1-2 tablets PO q4h PRN will be given. The number of tablets prescribed will depend on the extent of surgical trauma, as per a previously conducted study. As part of the standardized prescription group, patients will receive a handout (encouraging them to use non-opioid analgesics along with the opioid prescription to minimize their narcotic consumption).

Participants will be asked a series of questions via telephone consultation or in the pre-operative waiting area about their current opioid use, as well as their risk for narcotic abuse using the opioid risk tool (ORT). Participants will also be asked to fill out questionnaires assessing components of neuropathic pain (DN-4), any elements of anxiety or depression (HADS), and any tendencies for catastrophizing (PCS).

At the time of discharge participants will then be provided with either the standardized prescription or the usual discharge prescription by the surgeon.

Patients will be called after discharge from hospital on post-discharge weeks 1, 6, and 12 by either clinical investigators or research assistants. Patients will be asked standardized questions about their pain with the goal of assessing our primary endpoint of number of opioid pills used as compared to number prescribed. Patients will be attempted to be reached by telephone up to 3 times during the 7 day period following each pre-defined time point (i.e. 1, 6 and 12 weeks).

Subsequently the proportion of unused opioid pills will be calculated for each group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting to TWH for elective ambulatory hand and forearm surgery

Exclusion Criteria:

1. Chronic opioid treatment, defined as more than 6 tablets of Oxycodone 5 mg per day (or equivalent)
2. Cognitive impairment or any other condition causing inability to use 'as required' medication for pain control
3. Language barrier preventing completion of patient diary
4. Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of Standardized prescription on quality of analgesia after hand and forearm surgery | Twelve weeks after intervention

SECONDARY OUTCOMES:
Incidence of adverse effects of opioid medications experienced by patients | One week, Six weeks and Twelve weeks after intervention
Correlation of opioid consumption to pain scores | One week, Six weeks and Twelve weeks after intervention
Correlation of opioid consumption to functional limitations post-operatively as measured by the Disabilities of Arm Shoulder and Hand (DASH) score | Six weeks and Twelve weeks after intervention compared to pre-intervention
Incidence of disposal practices of prescribed opioids by patients | One week, Six weeks and Twelve weeks after intervention
  To indicate the type and incidence of disposal practices of prescribed opioids for patients (returned to pharmacy, retaining pills at home, and self-disposal of medication by participants
Patient satisfaction with pain management after discharge (as measured on a 0 to 10 scale, 0 being completely dissatisfied, and 10 being completely satisfied) | One week, Six weeks and Twelve weeks after intervention
The mean number of days patients require post-discharge opioid medications | One week, Six weeks and Twelve weeks after intervention
The correlation between in-hospital opioid analgesic requirements and post-discharge opioid consumption (all converted to oral morphine equivalents) | One week, Six weeks and Twelve weeks after intervention
The proportion of patients that require additional opioid prescription(s), on top of what is given at discharge, during the follow-up period, and 12 weeks | One week, Six weeks and Twelve weeks after intervention
The incidence of neuropathic pain as diagnosed by DN4 score >3/10 | Twelve weeks after intervention compared to pre-intervention
Impact of Standardized prescription on quality of analgesia after hand and forearm surgery | One week after intervention
Impact of Standardized prescription on number of unused opioid medications after hand and forearm surgery | One week after intervention
Impact of Standardized prescription on quality of analgesia after hand and forearm surgery | Six weeks after intervention
Impact of Standardized prescription on number of unused opioid medications after hand and forearm surgery | Six weeks after intervention

OTHER OUTCOMES:
Correlation of patient anxiety on pain numerical rating scores (0-10) | Twelve weeks after intervention compared to pre-intervention
Correlation of patient anxiety on opioid consumption | Twelve weeks after intervention compared to pre-intervention
Correlation of patient depression on pain numerical rating scores (0-10) | Twelve weeks after intervention compared to pre-intervention
Correlation of patient depression on opioid consumption | Twelve weeks after intervention compared to pre-intervention
Correlation of patient catastrophizing on pain numerical rating scores (0-10) | Twelve weeks after intervention compared to pre-intervention
Correlation of patient catastrophizing on opioid consumption | Twelve weeks after intervention compared to pre-intervention
Correlation of patient's score on the opioid risk tool (ORT) on post-op opioid use | Twelve weeks after intervention compared to pre-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, MD FRCPC, Principal Investigator — UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No